CLINICAL TRIAL: NCT00184015
Title: Bortezomib and Bevacizumab ("BB-mib-mab") in Patients With Advanced or Recurrent Renal Cell Cancer (RCC)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4K-05-1
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; Bortezomib

ARMS (2):
- Schedule A (Experimental)
  Interventions: Drug: Bevacizumab and Bortezomib
- Schedule B (Experimental)
  Interventions: Drug: Bevacizumab and Bortezomib

INTERVENTIONS:
Drug: Bevacizumab and Bortezomib — Bevacizumab 15 mg/kg on day 1 with Bortezomib 1.0 or 1.3 mg/m2 on days 1, 4, 8 and 11 every 21 days
  Arms: Schedule A
Drug: Bevacizumab and Bortezomib — Bevacizumab 15 mg/kg on day 1 with Bortezomib 1.6 or 1.8 mg/m2 on days 1 and 8 every 21 days
  Arms: Schedule B

SUMMARY:
This research study is for subjects with cancer of the kidney (also known as renal cell carcinoma) that cannot be treated with surgery. The purpose of this study is to see if the combination of bevacizumab and bortezomib is safe and tolerable and can help people with kidney cancer. The investigators would also like to find out what dose of the study drugs can be used safely and effectively, whether the combination of these two drugs can decrease cancer symptoms and stop tumor growth, and how frequently serious side effects might occur with this combination.

The study will be conducted in two phases-Phase 1 and Phase 2. In Phase 1, subjects will be assigned to a fixed dose of bevacizumab and different strengths of bortezomib given at 2 different schedules. Phase 2 will depend on how subjects tolerate the doses and schedules of bortezomib in Phase 1.

Bortezomib is a type of drug known as a "proteasome inhibitor." By blocking the "proteasome" in cancer cells, bortezomib affects the way these cells divide. Bevacizumab is an inhibitor (blocker) of blood vessel formation. Tumors need blood vessels in order to continue to grow and bevacizumab is thought to work by preventing new blood vessels from growing.

Bortezomib (also called Velcade or PS-341) has been approved by the US Food and Drug Administration (FDA) for the treatment of myeloma, but has not been approved for the treatment of kidney cancer. Bevacizumab (also called Avastin) has been approved by the FDA for the treatment of colon cancer, but has not been approved for the treatment of kidney cancer. However, the FDA is permitting the combined use of bortezomib and bevacizumab in this research study.

The bevacizumab that will be given in this study is not a commercially marketed product. Although it is expected to be very similar in safety and activity to the commercially available drug, it is possible that some differences may exist. Because this is not a commercially marketed drug, bevacizumab can only be administered to subjects enrolled in this study and may only be administered under the direction of physicians who are investigators in this study.

Approximately 40-52 subjects will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* Distant metastatic (TX NX M1) or locally recurrent renal cell carcinoma not amenable to cure by surgical or other means
* Measurable or non-measurable (evaluable) disease either on imaging scan or physical examination
* Pathological confirmation of the diagnosis of renal cell carcinoma either during prior nephrectomy or by biopsy of a primary or metastatic lesion - provision of a paraffin-embedded tissue block to confirm the diagnosis and allow molecular correlate assessment is required.
* ECOG performance status 0 or 1.
* Patients must have an AGC of greater than or equal to 1,500/mm3 and a platelet count of greater than or equal to 100,000/mm3. These tests must be obtained within 28 days of registration.
* Patients must have a calculated or measured creatinine clearance greater than or equal to 40 ml/min obtained within 28 days prior to registration.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method of contraception for the duration of the study.
* May have been treated with interleukin and/or interferon but must not have had more than one line of prior cytotoxic chemotherapy
* May have had up to one biologic therapy provided they have not had bortezomib or bevacizumab
* May have had up to 2 prior vaccine therapies
* May have been treated with radiation therapy, provided there are measurable or evaluable lesions outside the field of radiation
* May have had radiation provided the patient has recovered from the side effects of the therapy (typically 2 weeks after final fraction) and less than 30% of the total bone marrow has been irradiated

Exclusion Criteria:

* Brain metastases or history of brain metastases
* History of deep vein thrombosis or thromboembolic disease within 1 year or requiring ongoing anticoagulant therapy
* History of stroke or myocardial infarction within six months
* Other major illnesses likely to limit survival including poorly controlled hypertension (BP > 150/100 mmHg) or symptomatic or clinically significant peripheral vascular disease or angina pectoris
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* Urine protein:creatinine ratio greater than or equal to 1.0 at screening
* Evidence of bleeding diathesis or coagulopathy.
* Major surgical procedure, open biopsy, significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 0
* Pregnant (positive pregnancy test) or lactating; confirmation that female subject is not pregnant by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Inability to comply with study and/or follow-up procedures
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Neuropathy at baseline > grade 1
* Patient has received other investigational drugs within 14 days before enrollment
* Patient has hypersensitivity to bevacizumab, bortezomib, boron or mannitol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-08-18 (Actual); Primary Completion 2016-08-21 (Actual); Study Completion 2018-08-21 (Estimated)

PRIMARY OUTCOMES:
Toxicity | Toxicity as assessed by CTCAE 3.0 undertaken every 3 weeks

SECONDARY OUTCOMES:
response | Every 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Quinn, MD, PhD, Principal Investigator — University of Southern California
Locations (1):
- Norris Comprehensive Cancer Center, Los Angeles, California, United States